CLINICAL TRIAL: NCT01794910
Title: A Randomized Controlled Trial Comparing the Effect of Pelvic Floor Muscle Training on Improving Muscle Strength of Women After Vaginal or Cesarean Delivery
Brief Title: A Randomized Controlled Trial Comparing the Effect of Pelvic Floor Muscle Training
Acronym: PFMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Federal University of Maranhao (Other)
Responsible Party: Principal Investigator, LUIZ GUSTAVO OLIVEIRA BRITO, Assistant Physician, Department of Gynecology and Obstetrics, Ribeirao Preto School of Medicine, Sao Paulo University, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1136-5605
Record Dates: First submitted 2013-02-07; First posted 2013-02-20 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Pelvic Floor Muscle Weakness
Keywords: Pregnancy; Pelvic Floor; Muscle strength; Exercise therapy; natural childbirth; cesarean section; physiotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plevic floor muscle therapy (Experimental): The pelvic floor muscle therapy to women with vaginal or cesarean deliveries involved perineal contraction exercises in the dorsal decubitus, sitting, and standing positions and was applied twice per week for a total of 15 sessions.
  Interventions: Other: Pelvic floor muscle therapy
- Controll group (No Intervention): Women with vaginal or cesarean deliveries did not did not undergo muscle training

INTERVENTIONS:
Other: Pelvic floor muscle therapy — The women performed perineal contraction exercises in the dorsal decubitus, sitting, and standing positions and was applied twice per week for a total of 15 sessions
  Arms: Plevic floor muscle therapy

SUMMARY:
Aim: To determine the effects of pelvic floor muscle training (PFMT) in women with a single delivery route. Pregnancy and delivery route alter the pelvic floor muscle strength and are considered risk factors for urinary incontinence and genital dystopias. Methods: A Randomized controlled clinical trial with two hundred ninety-seven women aged 35 to 45 years old were selected for functional assessments of their pelvic floors by vaginal digital palpation and perineometry. One hundred sixty-five (69.7%) exhibited muscle strength deficits and were included in the clinical trial. The participants were distributed into two groups based on the delivery route (A, vaginal delivery and B, cesarean delivery) and were then randomly subdivided into Groups A1 (n = 44) and B1 (n = 42), who performed PFMT, and Groups A2 (n = 39) and B2 (n = 40), who did not undergo muscle training. The PFMT involved perineal contraction exercises in the dorsal decubitus, sitting, and standing positions and was applied twice per week for a total of 15 sessions. The functional assessment of pelvic floor by vaginal digital palpation and perineometry was performed after 15 sessions of pelvic´s floor muscles training. The statistical analysis was performed using the Mann-Whitney and Z tests at a 5% level of significance.

ELIGIBILITY:
Inclusion Criteria:

* age between 35 and 45 years old, obstetric antecedent of a single delivery route (i.e., vaginal or abdominal), and regular menstrual cycles for six months prior to the initial interview.

Exclusion Criteria:

* women who had complaints or clinical manifestations suggestive of urinary incontinence, intense pelvic or vaginal pain, past histories of physical therapy for pelvic floor strengthening, correction of genital prolapse, myomectomy, (total or subtotal) hysterectomy, morbidities such as diabetes and arterial hypertension, or body mass indices (BMIs) that were determined during the physical examination to be equal to or higher than 30 kg/m2.

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 297 (Actual)
Dates: Start 2010-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Pelvic floor muscle strength by two methods | The strength of pelvic floor muscle by digital palpation and perineometry were evaluated one day after 15 sessions of pelvic floor muscle training.
  Verification of pelvic floor muscle strength by digital palpation and perineometry before application of exercise and after 15 visits

SECONDARY OUTCOMES:
Application of a questionnaire | One day after 15 sessions of pelvic floor muscle training.
  Verification of age,type of delivery, number of deliveries through a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Maria Bethânia C Chein, phD, Study Director — Federal University of Maranhao
Locations (1):
- Post Graduate Program of Maternal and Child Health, São Luís, Maranhão, Brazil